CLINICAL TRIAL: NCT00786864
Title: School-Based Specific Exercise Programme Reduces the Prevalence and Intensity of Low Back Pain in 12-13 Year Old Children: a Randomized Controlled Trial
Brief Title: Exercise for Low Back Pain in Children
Acronym: LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Gina Lucia Fanucchi, University of the Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Fanucchi et al; M060334
Record Dates: First submitted 2008-10-14; First posted 2008-11-06 (Estimated); Results first posted 2008-11-06 (Estimated); Last update posted 2008-11-06 (Estimated); Status verified 2008-11

CONDITIONS: Low Back Pain
Keywords: Randomised controlled trial; low back pain; exercise; children; school-based; prevalence; intensity
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Experimental Group (Experimental): Exercise Intervention Group
  Interventions: Other: exercise programme
- 2. Control Group (No Intervention): Control group - no intervention

INTERVENTIONS:
Other: exercise programme — Specific low back pain exercise programme for children
  Arms: 1. Experimental Group

SUMMARY:
This study aimed to determine the efficacy of an eight-week specific exercise programme in reducing self-reported episodes and intensity of LBP, as well as modifying some of the identified risk factors for LBP, in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-13 years
* Complained of LBP in the past three months

Exclusion Criteria:

* Serious spinal pathologies or deformities (e.g. severe scoliosis, spinal tumours)
* Neurological conditions which alter motor tone
* Physical disabilities (e.g. spinal cord injuries) which prevent the child from being able to stand up on their own without an orthotic device or brace, or which prevent the child from taking part in normal physical education (PE) classes
* Any other serious co-morbidities (e.g. cancer, severe lung pathology)
* Provincial sports participants, or children who were currently following a specific training programme with a biokineticist or physiotherapist
* Current orthopaedic procedures or fractures of the spine, pelvis, lower or upper limbs

Ages: 12 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina L Fanucchi, MSc (Physio), Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Government primary schools in the Ekurhuleni West and Johannesburg East Districts of Gauteng, Johannesburg, Gauteng, South Africa

REFERENCES:
- [Derived] Fanucchi GL, Stewart A, Jordaan R, Becker P. Exercise reduces the intensity and prevalence of low back pain in 12-13 year old children: a randomised trial. Aust J Physiother. 2009;55(2):97-104. doi: 10.1016/s0004-9514(09)70039-x. PMID 19463080

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited January 2007 from 2 Government primary schools in the Ekurhuleni West and Johannesburg East Districts of Gauteng
Pre-assignment Details: Only children who met the inclusion criteria for the study were included
Groups:
- Exercise Intervention Group: Experimental Group
- Control Group: Control group - no intervention
Period: Overall Study
Arm/Group | Exercise Intervention Group | Control Group
Started | 39 | 33
Completed | 38 (1 child excluded at the 3 month follow-up, as he sustained a serious back injury) | 32 (1 child lost to study immediately post-intervention as she left the school)
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Sustained serious back injury | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Intervention Group | Control Group | Total
Number analyzed (Participants) | 39 | 33 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 39 | 33 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12.21 (0.66) | 12.39 (0.70) | 12.29 (0.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 15 | 39
  Male | 15 | 18 | 33
Region of Enrollment [Number; unit: participants]
  South Africa | 39 | 33 | 72

OUTCOME MEASURES:

1. Primary Outcome: Low Back Pain Prevalence
Description: All of the children complained of low back pain at baseline. Low back pain prevalence post-intervention was determined by the number of children still complaining of low back pain post-intervention.
Time Frame: 3 months post-intervention
Population: Intention to treat analysis
Measure: Number; unit: participants
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 38 | 32
participants | 16 | 26
Statistical Analysis 1: Comparison: Exercise Intervention Group vs Control Group; Test type: Superiority or Other; p = 0.001, ANCOVA

2. Secondary Outcome: Neural Mobility
Description: Straight leg raise test was used to measure neural mobility. The amount of hip flexion (angle between the plinth and femur of the raised leg) was measured using a digital inclinometer. Scores ranged between 3 (worst score) and 90.5 (best score). Continuous data.
Time Frame: 3 months post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 38 | 32
degrees | 64.41 (17.10) | 44.44 (16.55)
Statistical Analysis 1: Comparison: Exercise Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.001, ANCOVA

3. Primary Outcome: Low Back Pain Intensity
Description: The visual analogue scale (standardised 100mm, non-hatched line) was used to determine pain intensity. Scores can range between 0 and 10, with the worst possible pain/score = 10 and no pain/best score = 0. Visual analogue scale is continuous.
Time Frame: 3 months post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 38 | 32
units on a scale | 1.76 (2.59) | 3.73 (3.06)
Statistical Analysis 1: Comparison: Exercise Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.001, ANCOVA

4. Secondary Outcome: Hamstring Flexibility
Description: Standardised hamstring muscle length test. The child was positioned in supine, with the hip flexed at 90 degrees. The knee was then extended passively. The angle of knee extension [from horizontal plane (level to plinth) to fibula] was measured using a digital inclinometer. Continuous data. Scores ranged from -20 (worst score) to 82 (best score).
Time Frame: 3 months post-intervention
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Exercise Intervention Group | Control Group
Number analyzed (Participants) | 38 | 32
degrees | 54.00 (11.87) | 45.76 (9.59)
Statistical Analysis 1: Comparison: Exercise Intervention Group vs Control Group; Test type: Superiority or Other; p < 0.01, ANCOVA

ADVERSE EVENTS:
Arm/Group | Exercise Intervention Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0 | 0
Other Adverse Events (participants affected / at risk) | 0 | 0

LIMITATIONS AND CAVEATS:
Only 2 schools, in a similar geographic and socioeconomic area were included, and therefore the results may not necessarily be generalized to a larger population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No